CLINICAL TRIAL: NCT00246701
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Combined Omacor and Simvastatin Therapy in Hypertriglyceridemic Subjects
Brief Title: Evaluation of Efficacy and Safety of Combined Omacor (Omega-3-acid Ethyl Esters) and Simvastatin Therapy in Hypertriglyceridemic Subjects
Acronym: COMBOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OM6 program (Reliant); LOV111818 (Other: GSK)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hypertriglyceridemia
Keywords: omega-3-acid ethyl esters; simvastatin; Lovaza; High triglycerides
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Simvastatin; Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Active Comparator): Simvastatin + placebo
  Interventions: Drug: Simvastatin
- Simvastatin + Lovaza (Experimental): Simvastatin + Lovaza (omega-3-acid ethyl esters)
  Interventions: Drug: Simvastatin + Lovaza

INTERVENTIONS:
Drug: Simvastatin — Simvastatin
  Arms: Simvastatin
Drug: Simvastatin + Lovaza — Simvastatin + Lovaza (omega-3-acid ethyl esters)
  Arms: Simvastatin + Lovaza

SUMMARY:
The purpose of OM6 is to evaluate efficacy and safety of Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor] combined with simvastatin for lowering non-high-density lipoprotein cholesterol (non-HDL-C) in subjects with persistent high triglycerides despite statin therapy.

Additionally, a two-year extension trial (LOV111818/OM6X) is posted on NCT00903409.

DETAILED DESCRIPTION:
Two studies comprise this OM6 Program. Study OM6 / LOV111858 (double-blind study) and is not required to post results based on FDAAA. Study OM6X / LOV111818 (open-label extension) is posted on NCT00903409.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-79 years, inclusive
* Current therapy with a statin drug
* Triglyceride levels between 200 and 499 mg/dL
* Normally active and in good health on the basis of medical history, brief physical examination, electrocardiogram, and routine laboratory tests
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Sensitivity to statin drugs or omega-3 fatty acids
* Lipoprotein lipase impairment or apo C-2 deficiency or type III hyperlipidemia
* Unexplained muscle pain or weakness
* History of pancreatitis
* Recent history of certain heart, kidney, liver, lung, or gastrointestinal diseases, or cancer (except non-melanoma skin cancer)
* Poorly controlled diabetes, or receiving insulin therapy
* Pregnant or lactating females. Women of childbearing potential who are not using a medically approved method of contraception.
* Use of certain types of hormones, anticonvulsant drugs, immunologic drugs, antibiotic, antifungal and antiviral drugs, and cardiac drugs
* Use of warfarin (Coumadin)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2005-11-01 (Actual); Primary Completion 2006-06-01 (Actual); Study Completion 2006-06-01 (Actual)

PRIMARY OUTCOMES:
Difference between simvastatin + Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor] and simvastatin + placebo treatment groups in the percent change from baseline to end-of-treatment in non-high-density lipoprotein cholesterol | 8 weeks

SECONDARY OUTCOMES:
OM6/LOV111858 - Difference between simvastatin + Lovaza (omega-3-acid ethyl esters) and simvastatin + placebo treatment groups in the percent change from baseline to end-of-treatment in other lipid and biomarker levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Maki KC, Dicklin MR, Davidson MH, Doyle RT, Ballantyne CM; COMBination of prescription Omega-3 with Simvastatin (COMBOS) Investigators. Baseline lipoprotein lipids and low-density lipoprotein cholesterol response to prescription omega-3 acid ethyl ester added to Simvastatin therapy. Am J Cardiol. 2010 May 15;105(10):1409-12. doi: 10.1016/j.amjcard.2009.12.063. Epub 2010 Mar 30. PMID 20451686